CLINICAL TRIAL: NCT02936206
Title: Comparison in the Change of Proliferation Index Between Fulvestrant and Tamoxifen in Cyclin D1 +, Estrogen Receptor + Breast Cancer
Brief Title: Examination of Breast Cancer Cells of Pre-menopausal and Post-menopausal Women Before and After Exposure to Tamoxifen or Fulvestrant.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual rate
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Amy Tiersten, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GCO 16-1470
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Results first posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
Keywords: proliferation Index; Tamoxifen; Fulvestrant; cyclinD1; Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fulvestrant (Experimental): 750 mg injection in 3 divided doses
  Interventions: Drug: Fulvestrant
- Tamoxifen (Active Comparator): 20mg orally
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Fulvestrant — fulvestrant 750 mg (three 5 ml injections slowly over 1-2 mn per injection in the buttocks) on day 1 only
  Other Names: Faslodex
  Arms: Fulvestrant
Drug: Tamoxifen — 14 days of treatment with tamoxifen 20mg orally each day
  Other Names: Nolvadex
  Arms: Tamoxifen

SUMMARY:
The purpose of this study is to microscopically examine breast cancer cells of pre-menopausal and post-menopausal women before and after exposure to one of the two commonly used breast cancer drugs, tamoxifen or fulvestrant.

DETAILED DESCRIPTION:
The researchers hypothesize that the cyclinD1-interactome can be used to orient the use of fulvestrant in premenopausal and postmenopausal women. To test this hypothesis, the researchers propose a pre-surgical randomized clinical trial of tamoxifen vs fulvestrant in the window between breast cancer diagnosis on core biopsy and definitive surgery. Women with ER/cyclinD1 positive tumors will be eligible. Response to tamoxifen or fulvestrant will be evaluated using standard proliferation index as well as gene expression signatures obtained in pre-clinical models of tamoxifen resistance and sensitivity to fulvestrant. In addition, the researchers propose to use cutting edge new technology allowing ex-vivo expansion of primary culture from only a few cancer cells obtained by fine needle biopsy. The researchers propose to compare the response of these primary cells to patient response. If successful, the impact of this work can support the expansion of use of fulvestrant to not only postmenopausal women but premenopausal women as well. In addition, it may serve as a proof of principle to maximize the use of biopsy material to predict treatment response

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the patients for the study treatment regimen and follow-up, must be obtained and documented according to the local regulatory requirements
* Adult women greater than 18 years old
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* New diagnosis of invasive cyclin D1 +, ER+, PR +/-, Her2- breast cancer

  * Cyclin D1 positive as defined as a total immunohistochemical score of 5 or greater
  * Hormone receptor positive as defined as ≥ 10% positive stained cells
  * HER2-normal (IHC score 0-1 or FISH negative [in-situ hybridization (ISH) ratio <= 2.0 status])
* Tumor size at least 5 mm with planned primary surgery at Mount Sinai
* A negative urine dipstick pregnancy test

Exclusion Criteria:

* Estrogen receptor negative invasive breast carcinoma as defined as less than 10% stained cells
* Prior antiestrogen therapy
* Tumor size less than 5 mm
* Prior diagnosis of thrombosis or known hypercoagulable state
* Known history of bleeding diathesis
* Known liver disease
* Prior treatment with neoadjuvant therapy
* Inflammatory breast cancer defined as clinically significant erythema of the breast and/or documented dermal lymphatic invasion (not direct skin invasion by tumor or peau d'orange without erythema).
* Current severe or uncontrolled systemic disease
* Pregnancy or lactation period. Patients of childbearing potential must implement adequate non-hormonal contraceptive measures (barrier methods, intrauterine contraceptive devices) during study treatment.
* Prior malignancy (including invasive or ductal in-situ breast cancer) within 5 years prior to randomization, except curatively treated basal cell carcinoma of the skin and carcinoma in situ of the cervix.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-10; Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Tiersten, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Mount Sinai West, New York, New York
  - Mount Sinai St. Luke's, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fulvestrant | Tamoxifen
Started | 0 | 2
Completed | 0 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were 2 participants in the study, both randomized to Tamoxifen arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fulvestrant | Tamoxifen | Total
Number analyzed (Participants) | 0 | 2 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 2 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Ki67 Cell Percentage
Description: The change in proliferation index as measured by the percentage of cells staining for Ki67 at 2 weeks as compared on baseline.
Time Frame: baseline and 2 weeks
Population: With the 2 patients enrolled on the trial, the data collected was insufficient and not evaluable.
Arm/Group | Fulvestrant | Tamoxifen
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Estrogen Receptor Level
Description: The change in estrogen receptor level at 2 weeks as compared to baseline.
Time Frame: baseline and 2 weeks
Population: With the 2 patients enrolled on the trial, the data collected was insufficient and not evaluable.
Arm/Group | Fulvestrant | Tamoxifen
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Progesterone Receptor Level
Description: The change in progesterone receptor level at 2 weeks as compared to baseline.
Time Frame: baseline and 2 weeks
Population: With the 2 patients enrolled on the trial, the data collected was insufficient and not evaluable.
Arm/Group | Fulvestrant | Tamoxifen
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Incidence of Tamoxifen-resistance Gene Expression
Description: Number of tamoxifen-resistance gene expression signature observed in patients with cyclinD1 overexpressing breast cancers.
Time Frame: 2 weeks
Population: With the 2 patients enrolled on the trial, the data collected was insufficient and not evaluable.
Arm/Group | Fulvestrant | Tamoxifen
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Incidence of Fulvestrant-sensitivity Gene Expression
Description: Number of fulvestrant-sensitivity gene expression signature observed in patients with cyclinD1 overexpressing breast cancers.
Time Frame: 2 weeks
Population: With the 2 patients enrolled on the trial, the data collected was insufficient and not evaluable.
Arm/Group | Fulvestrant | Tamoxifen
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Drug Dose Level
Description: For samples that are available for culture in vivo, proliferation assay to test whether the cells derived from individual patients respond the same as the tumor in vivo in the same patient.
Time Frame: 2 weeks
Population: With the 2 patients enrolled on the trial, the data collected was insufficient and not evaluable.
Arm/Group | Fulvestrant | Tamoxifen
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Cells Staining Positive Within the Breast Tumor
Description: Differential treatment effect for pre and post menopausal subjects assessed by the mean change in levels (expressed as a percentage of cells staining positive within the breast tumor) of ER (and PR) between pre-treatment and post-treatment stratified by menopausal status.
Time Frame: 2 weeks
Population: With the 2 patients enrolled on the trial, the data collected was insufficient and not evaluable.
Arm/Group | Fulvestrant | Tamoxifen
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: not collected
Description: not collected
Arm/Group | Fulvestrant | Tamoxifen
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT02936206/Prot_SAP_000.pdf